CLINICAL TRIAL: NCT03724032
Title: Investigation and Modulation of the Mu-opioid Mechanisms in TMD (in Vivo)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Alexandre DaSilva, DDS, DMedSc, Associate Professor, BMS-Prosthodontics Dept., School of Dentistry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00110179; U01DE025633 (NIH)
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- TMD Patients Active Group: Active Comparator (Active Comparator): 30 TMD patients will be randomized (Taves method) to receive high-definition transcranial direct current stimulation (HD-tDCS*) as 20 minute sessions, once daily for 10 days (M-F for 2 weeks).
  Interventions: Device: HD-tDCS*
- TMD Patients Sham Group: Sham Comparator (Sham Comparator): 30 TMD patients will be randomized (Taves method) to receive high-definition transcranial direct current stimulation (HD-tDCS*) as 30-second administrations at the beginning and end of each 20 minute session, once daily for 10 days (M-F for 2 weeks).
  Interventions: Device: Sham HD-tDCS*
- Healthy Control Group (No Intervention): 20 Healthy Volunteers will be asked to undergo baseline assessments only (including imaging, but no brain stimulation).
  Healthy volunteer data (n </= 10) may be used from a prior study (NIDCR-R56-DE022637 project [IRBMED #HUM00080911; Dr. Alexandre DaSilva, Principal Investigator]). Consent to use data for a future study was obtained in the informed consent document at the time of participation.

INTERVENTIONS:
Device: HD-tDCS* — Non-invasive brain stimulation (active protocol)
  Other Names: HD-tDCS (active protocol)
  Arms: TMD Patients Active Group: Active Comparator
Device: Sham HD-tDCS* — Non-invasive brain stimulation (sham protocol)
  Other Names: HD-tDCS (sham protocol)
  Arms: TMD Patients Sham Group: Sham Comparator

SUMMARY:
In this study, this team of researchers will investigate the impact of chronic temporomandibular disorder suffering on the endogenous μ-opioid system in vivo, arguably one of the principal endogenous pain modulatory systems in the brain, and its modulation by 10 daily sessions of primary motor cortex stimulation using high-definition transcranial direct current stimulation (HD-tDCS).

DETAILED DESCRIPTION:
Approximately 10% of TMD patients will not experience an improvement of their symptoms and around 75% of patients who fail to respond to conservative treatments are also not suitable for TM joint surgery. Initial studies from NIH-NIDCR R56 project using positron emission tomography (PET) with [11C] Carfentanil, a selective radiotracer for μ-opioid receptor (μOR), have demonstrated that there is a decrease in thalamic μOR availability (non displaceable binding potential BPND) in the brains of TMD patients during masseteric pain compared to healthy controls. μ-opioid neurotransmission is arguably one of the mechanisms most centrally involved in pain regulation and experience. Moreover, the thalamus is the major relay structure in the forebrain for (non)-noxious inputs, which will be distributed subsequently to multiple cortical areas for discriminative, cognitive and affective processing. MRI-based reports have found that those findings co-localize with neuroplastic changes in trigeminal pain patients. Conventional therapies are unable to selectively target the thalamus and associated regions, and there is a paucity of data on how to reverse neuroplastic molecular mechanisms when available medications fail. Interestingly, several studies with motor cortex stimulation (MCS) have shown that epidural electrodes in the primary motor cortex (M1) are effective in providing analgesia in patients with central pain and that it occurs via indirect modulation of thalamic activity. Evidently, the invasive nature of such a procedure limits its indication to highly severe pain disorders. New non-invasive neuromodulatory methods for M1, such as transcranial direct current stimulation (tDCS), can now safely modulate the μOR system, providing relatively lasting pain relief in pain patients. Recently, a novel high-definition tDCS (HD-tDCS) montage created by this research group was able to reduce exclusively "contralateral" sensory-discrimative clinical pain measures (intensity/area) in TMD patients by targeting precisely the M1 region. Therefore, the main goals of this study are: First, to exploit the μ-opioidergic dysfunction in vivo in TMD patients compared to healthy controls; Second, to determine whether 10 daily sessions of noninvasive and precise M1 HD-tDCS have a modulatory effect on clinical and experimental pain measures in TMD patients; and Third, to investigate whether repetitive active M1 HD-tDCS induces/reverts μOR BPND changes in the thalamus and other pain-related regions, and whether those changes are correlated with TMD pain measures. The studies above represent a change in paradigm in TMD research, as this research group directly investigates and modulates in vivo one of the most important endogenous analgesic mechanisms in the brain.

The IRB approved study protocol also includes secondary data sets to be used for analysis in study objective #6 only. The data sets are not part of the clinical trial as they were collected during a previous study (NIDCR-R56-DE022637 project [IRBMED #HUM00080911; Dr. Alexandre DaSilva, Principal Investigator]). Participants in HUM00080911 (both Healthy and TMD patients) received no intervention, but underwent the same Baseline, MRI and PET protocol. This secondary data will not be represented in the Adverse Event or final enrollment total for this clinical trial. However, the data will be analyzed in a meta-analysis addressing secondary objective #6 only. These data sets will not be used to analyze any primary study objectives, nor change the terms of the clinical trial. Manuscripts that include these secondary data sets will clearly indicate the use of this data and clarify that the data was collected separate from the clinical trial data.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form;
* Male or female, aged 18 to 65 (inclusive);
* tDCS naïve; and
* Willing to comply with all study procedures and be available for the duration of the study.

In addition, TMD subjects must qualify as:

• Diagnosed with chronic TMD as defined by the Diagnostic Criteria (DC) for TMD and the American Academy of Orofacial Pain (DC/TMD): "Chronic TMD pain and dysfunction for at least one year from the clinical exam session (DC/TMD: Masticatory myofacial pain with/without referral) not adequately controlled by previous therapies (eg, NSAIDs, muscle relaxants)"

* TMJ open-surgery naïve;
* TMD maximum pain score pain of greater than or equal to 3 (moderate to severe) on a 0-10 VAS, despite existing treatment, for 3 days in the 7 days preceding study consent, based on report at the screening session;
* If taking pain medications, the dose regimen must be stable for at least 4 weeks prior to screening; and
* Willing to halt the introduction of new medications for chronic TMD symptoms during the study.

Emphasis is therefore placed on generalizability and chronicity of symptoms.

OR

To qualify as a Healthy Volunteer, subjects must be:

* Without self-reported history of systemic disorders or other chronic pain disorders, including migraine.

Exclusion Criteria:

* Existence of chronic pain disorder(s) other than TMD
* History of a traumatic brain injury
* History or current evidence of a psychotic disorder (e.g. schizophrenia) or substance abuse (self-reported)
* Bipolar or severe major depression, as evidenced by a Beck Depression Inventory score of ≥ 30
* Ongoing, unresolved disability litigation (self-reported)
* History of neurological disorder (e.g. epilepsy, stroke, neuropathy, neuropathic pain; self-reported)
* Opioid pain medications taken within the past 3 months
* Past allergic response to opioids or chemically related drugs (e.g., carfentanil)
* Excluded by MRI Center or PET Center safety screening checklist (as administered by study staff)
* Drug test positive for opioid or recreational drug (e.g., cannabis) at the time of the PET scan visits
* Pregnant or lactating (negative urine pregnancy test must be available before any PET procedures are initiated)
* Treatment with an investigational drug, device or other intervention within 30 days of study enrollment
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study (e.g., medical condition, laboratory finding, physical exam finding, logistical complication).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre F DaSilva, DDS, DMedSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim DJ, Nascimento TD, Lim M, Danciu T, Zubieta JK, Scott PJH, Koeppe R, Kaciroti N, DaSilva AF. Exploring HD-tDCS Effect on mu-opioid Receptor and Pain Sensitivity in Temporomandibular Disorder: A Pilot Randomized Clinical Trial Study. J Pain. 2024 Apr;25(4):1070-1081. doi: 10.1016/j.jpain.2023.11.001. Epub 2023 Nov 11. PMID 37956741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled a total of 15 participants into the protocol. Secondary data from an additional 12 participants who participated in a prior study were also incorporated into the analysis for some secondary outcome measures as noted in the protocol section.
Pre-assignment Details: After consent to participate, subjects underwent evaluation to ensure eligibility into the study. Several patients screen failed at this stage of the study. Additional inclusion/exclusion criteria required by the sponsor were highly strict for our patient community and excluded the majority of volunteers who were pre-screened (490 total pre-screened).
Period: Overall Study
Arm/Group | TMD Patients Active Group: Active Comparator | TMD Patients Sham Group: Sham Comparator | Healthy Control Group
Started | 6 | 6 | 15 (3 participants were enrolled in the study. Secondary data from an additional 12 participants was analyzed during the data analysis phase.)
Completed | 3 | 4 | 14
Not Completed | 3 | 2 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Please note that the healthy control group incorporates secondary data from 12 participants who did not enroll in the study protocol. These 12 participants are not reflected in the enrollment total, though they are reflected in the Participant flow and baseline analysis population total for analysis purposes.
Groups:
- Total: Total of all reporting groups
Arm/Group | TMD Patients Active Group: Active Comparator | TMD Patients Sham Group: Sham Comparator | Healthy Control Group | Total
Number analyzed (Participants) | 3 | 4 | 14 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 14 | 21
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (6.2) | 30.4 (9.1) | 27.6 (8.2) | 28.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 12 | 17
  Male | 1 | 1 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 14 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 2 | 4 | 12 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 14 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Visual Analog Scale Pain Score From Baseline (Screening Day) to 4 Weeks After Completion of HD-tDCS Sessions (Follow Up #2).
Description: Change in clinical Visual Analog Scale pain score from baseline (Screening Day) to 4 weeks after completion of HD-tDCS sessions (Follow Up #2). Pain is measured on a scale of 1-10, with 10 being the worst.
Time Frame: Screening (Baseline), 4 Weeks after completion of HD-tDCS sessions
Population: 2 subjects were excluded from analysis due to IRB requirements related to one pain measure threshold.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TMD Patients Active Group: Active Comparator | TMD Patients Sham Group: Sham Comparator
Number analyzed (Participants) | 2 | 3
units on a scale | -0.5 [-0.7 to 0.6] | -1.6 [-5.4 to 2.2]

2. Secondary Outcome: Change in Clinical Visual Analog Scale Pain Score During Sustained Masseteric Pain Stress Challenge From Baseline PET (#1) Session to Follow-up PET (#2) Session, 1 Week After Completion of HD-tDCS Sessions.
Description: Change in clinical Visual Analog Scale pain score during sustained masseteric pain stress challenge from baseline PET (#1) session to follow-up PET (#2) session, 1 week after completion of HD-tDCS sessions.
Time Frame: Baseline, 1 Week after completion of HD-tDCS sessions
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TMD Patients Active Group: Active Comparator | TMD Patients Sham Group: Sham Comparator
Number analyzed (Participants) | 3 | 4
units on a scale | 0 [-2.5 to 2.5] | 0.2 [-0.7 to 1.0]

3. Secondary Outcome: Changes in GeoPain Measures (PAINS - Summation of Area and Intensity) From Baseline Daily Over the Treatment Period and Through Follow-up (4 Weeks After Completion of HD-tDCS Sessions).
Description: Short- and long-term changes in GeoPain measures (percentage of pain area extension in the head region, average of pain intensity in the affected region, and their summation, meaning percentage of combined pain area and intensity in the affected region) from baseline daily over the treatment period and through follow-up at 4 weeks after completion of HD-tDCS sessions).
Time Frame: Baseline to 4 weeks after completion of HD-tDCS sessions
Population: 2 subjects were excluded from analysis due to IRB requirements related to one pain measure threshold.
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | TMD Patients Active Group: Active Comparator | TMD Patients Sham Group: Sham Comparator
Number analyzed (Participants) | 2 | 3
percentage | -4.8 [-122.5 to 112.8] | -2.1 [-17.1 to 13.0]

4. Secondary Outcome: Difference in µOR BPND Levels of Thalamus From Baseline PET (#1) Session to Follow-up PET (#2) Session, 1 Week After Completion of HD-tDCS Sessions.
Description: The difference in µOR BPND levels (a measure of receptor availability) between Baseline PET #1 and PET (#2) in TMD patients (active vs sham treatment groups).
  The values indicate changes in the availability of mu-opioid receptors (µOR), referred to as the non-displaceable binding potential (BPND), which reflects the density or concentration of available µORs in a particular region of interest in the brain, specifically the left thalamus. These changes are assessed by conducting baseline positron emission tomography (PET) scans prior to treatment and follow-up PET scans one week after the completion of HD-tDCS sessions. During each PET scan, µOR measurements are taken during an early resting phase. A positive value indicates increased µOR availability following treatment, while a negative value indicates decreased availability after treatment.
Time Frame: Baseline to 1 Week after completion of HD-tDCS sessions.
Measure: Mean (95% Confidence Interval); unit: arbitrary units
Arm/Group | TMD Patients Active Group: Active Comparator | TMD Patients Sham Group: Sham Comparator
Number analyzed (Participants) | 3 | 4
arbitrary units | 0.05 [0.03 to 0.07] | -0.02 [-0.2 to 0.2]

5. Secondary Outcome: Change in Clinical Visual Analog Scale Pain Score at Rest From Baseline PET (#1) Session to Follow-up PET (#2) Session, 1 Week After Completion of HD-tDCS Sessions.
Description: Change in clinical Visual Analog Scale pain score at rest from baseline PET (#1) session to follow-up PET (#2) session, 1 week after completion of HD-tDCS sessions.
Time Frame: Baseline, 1 Week after completion of HD-tDCS sessions.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TMD Patients Active Group: Active Comparator | TMD Patients Sham Group: Sham Comparator
Number analyzed (Participants) | 3 | 4
units on a scale | -2.5 [-10.2 to 5.1] | 0.2 [-0.6 to 1.1]

6. Secondary Outcome: Difference in µOR BPND Levels at Rest During PET (#1) in Chronic TMD Patients as Compared to Healthy Subjects.
Description: The difference in µOR BPND levels (a measure of receptor availability) at rest (5-40 mins after radiotracer injection) during baseline PET in TMD patients as compared to healthy subjects.
  The values for each group the availability of mu-opioid receptors (µOR), referred to as the non-displaceable binding potential (BPND), which reflects the density or concentration of available µORs in a particular region of interest in the brain, specifically the left thalamus. It was assessed by conducting baseline positron emission tomography (PET) scans. The outcome measure 6 was taken during an early-resting (outcome 6)
Time Frame: During PET #1, at rest (5-40 mins after radiotracer injection)
Measure: Mean (95% Confidence Interval); unit: arbitrary units
Arm/Group | TMD Patients Active Group: Active Comparator | TMD Patients Sham Group: Sham Comparator | Healthy Control Group
Number analyzed (Participants) | 3 | 4 | 14
arbitrary units | 1.8 [0.7 to 2.9] | 1.5 [1.3 to 1.8] | 1.5 [1.4 to 1.6]

7. Secondary Outcome: Difference in µOR BPND Levels During Experimental Sustained Masseteric Pain Stress Challenge During PET (#1) in Chronic TMD Patients as Compared to Healthy Subjects
Description: Difference in µOR BPND levels (a measure of receptor availability) at experimental sustained masseteric pain stress challenge (45-90 mins after radiotracer injection) during baseline PET in TMD patients as compared to healthy subjects.
  The values for each group the availability of mu-opioid receptors (µOR), referred to as the non-displaceable binding potential (BPND), which reflects the density or concentration of available µORs in a particular region of interest in the brain, specifically the left thalamus. It was assessed by conducting baseline positron emission tomography (PET) scans. The outcome measure 7 was taken during a late pain stimulus (hypertonic saline infusion) phase.
Time Frame: PET (#1) during experimental sustained masseteric pain stress challenge (45-90 mins after radiotracer injection)
Measure: Mean (95% Confidence Interval); unit: arbitrary units
Arm/Group | TMD Patients Active Group: Active Comparator | TMD Patients Sham Group: Sham Comparator | Healthy Control Group
Number analyzed (Participants) | 3 | 4 | 14
arbitrary units | 1.7 [0.5 to 2.9] | 1.5 [1.2 to 1.8] | 1.5 [1.4 to 1.6]

ADVERSE EVENTS:
Time Frame: During the 2-weeks of HD-tDCS treatment
Description: Adverse Events were collected using a questionnaire that reflects common side effects of tDCS treatment. The questionnaire was administered before and after each of 10 tDCS treatment sessions. All of the adverse events reported were expected and mild in severity.
Groups:
- Active TMD Patients: TMD patients who received active HD-tDCS treatment for 10 days
- Sham TMD Patients: TMD patients who complete 10 sham treatments
- Healthy Volunteers: Healthy Volunteers did not receive treatment.
Arm/Group | Active TMD Patients | Sham TMD Patients | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/15
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active TMD Patients (N=4) | Sham TMD Patients (N=4) | Healthy Volunteers (N=15)
Headache (Investigations) | 3 | 1 | NA
Scalp Pain (Investigations) | 2 | 1 | NA
Scalp Burn sensation (mild) (Investigations) | 1 | 1 | NA
Tingling (Investigations) | 2 | 3 | NA
sleepiness (Investigations) | 2 | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT03724032/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03724032/ICF_001.pdf